CLINICAL TRIAL: NCT07223840
Title: A Phase 2, Multicenter, Randomized, Double-Blind Study to Investigate the Efficacy and Safety of Brenipatide Compared With Placebo for Reduction in Risk of Relapse to Cigarette Smoking in Adults (RENEW-Smk-1)
Brief Title: A Study of Brenipatide in Adults Who Quit Smoking Cigarettes and Want to Avoid Relapse
Acronym: RENEW-Smk-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27411; J2S-MC-GZMO (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-10-31; First posted 2025-11-03 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brenipatide (Experimental): Brenipatide administered subcutaneously (SC).
  Interventions: Drug: Brenipatide
- Placebo (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brenipatide — Administered SC
  Other Names: LY3537031
  Arms: Brenipatide
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy and safety of brenipatide when compared to placebo for reducing the risk of relapse to cigarette smoking in adults who have recently quit.

Study participation will last approximately 34 weeks with up to 17 study visits, which includes a 2-week screening period, 24-week treatment period, 8-week safety follow-up period.

.

ELIGIBILITY:
Inclusion Criteria:

* Have recently quit smoking and are motivated to stay quit from smoking
* Are reliable and willing to make themselves available for the duration of the study and attend required study visits and are willing and able to follow study procedures as required, such as self-inject study intervention

Exclusion Criteria:

* Have evidence of any substance use disorder within the past 180 days prior to screening, except mild alcohol use disorder, mild cannabis use disorder, or tobacco use disorder
* Have answered "yes" to either Question 4 or Question 5 on the "Suicidal Ideation" portion of the C-SSRS and the ideation occurred within the past 6 months, or have answered "yes" to any of the suicide-related behaviors on the "Suicidal Behavior" portion of the C-SSRS and the behavior occurred within the past 6 months
* Have severe chronic obstructive pulmonary disease, or any other clinically severe respiratory condition that in the investigator's opinion may pose a risk.
* Have participated in a clinical study and have received active treatment, or unknown if they received active treatment, within 90 days or 5 half-lives (whichever is longer) before screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants that Achieve Carbon Monoxide (CO)-Confirmed Continuous Abstinence from Cigarette Smoking with Allowed Slips | Week 1 to Week 24

SECONDARY OUTCOMES:
Number of Participants That Achieve CO-confirmed Continuous Abstinence from Cigarette Smoking Without Allowed Slips | Week 1 to Week 24
Mean Change from Baseline in Patient Reported Outcomes | Baseline, Week 24
Mean Percentage Change in Body Weight | Baseline, Week 24
Pharmacokinetic (PK): Average Steady State Plasma Concentration (Cavg) of Brenipatide | Baseline up to Week 24
Number of Treatment-emergent Anit-drug Antibodies | Baseline up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (28):
- United States (17):
  - Woodland Research Northwest, Rogers, Arkansas
  - Hillcrest Medical Research, DeLand, Florida
  - TecTum Research, Hollywood, Florida
  - K2 Medical Research ORLANDO, Maitland, Florida
  - GTL Medical & Research Group, Miami, Florida
  - North Georgia Clinical Research, Woodstock, Georgia
  - Revival Research Institute, LLC, Dearborn, Michigan
  - Arch Clinical Trials, St Louis, Missouri
  - Vector Clinical Trials, Las Vegas, Nevada
  - Rochester Clinical Research, LLC, Rochester, New York
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Circle Clinical Research, Sioux Falls, South Dakota
  - FutureSearch Trials of Dallas, Dallas, Texas
  - NextStage Clinical Research_Houston (07) -Menninger Clinic, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Eastside Research Associates, Redmond, Washington
- China (8):
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing
  - Beijing Anding Hospital - Affiliated Capital University of Medical Science, Beijing
  - Sichuan Provincial People's Hospital, Chengdu
  - 2nd Affiliated Hospital Chongqing Medical University, Chongqing
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou
  - Taizhou Hospital of Zhejiang Province, Linhai
  - The first affiliated hospital of Ningbo university, Ningbo
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen
- Japan (3):
  - Miyazaki RC Clinic, Shinagawa-ku
  - Samoncho Clinic, Shinjuku
  - Higashi Shinjuku Clinic, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal should be approved by an independent review panel and researchers should sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Brenipatide in Adults Who Quit Smoking Cigarettes and Want to Avoid Relapse (RENEW-Smk-1) — https://trials.lilly.com/en-US/trial/663855